CLINICAL TRIAL: NCT06116513
Title: Efficacy of Secondary Obliteration of Chronically Discharging Old Radical Cavities Using S53P4 Bioactive Glass
Brief Title: Secondary Obliteration of Old Radical Cavities Using S53P4 Bioactive Glass
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Diakonessenhuis, Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: 16-004-1
Record Dates: First submitted 2023-09-18; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Mastoid Cavity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with old troublesome radical cavities: These patients would have old Canal Wall Down cavities that were troublesome
  Interventions: Device: S53P4 bioactive glass granules

INTERVENTIONS:
Device: S53P4 bioactive glass granules — During revision surgery, all infectious material would be removed and subsequently the posterior wall of the external ear canal would be reconstructed and the mastoid would be obliterated using S53P4 bioactive glass.

SUMMARY:
In canal wall down surgeries, the posterior bony wall of the external auditory canal (EAC) is removed to increase exposure. The creation of a so-called radical cavity comes with several possible disadvantages, such as higher rates of postoperative otorrhea and purulence, pain, adherence to water precautions and dizziness. Secondary obliteration of the mastoid cavity and reconstruction of the posterior wall of the EAC can help alleviate these symptoms. Our goal is to study the efficacy of secondary obliteration using S53P4 bioactive glass as obliteration material. This bioactive glass has several important characteristics, such as retaining of volume over time and antibacterial effects. The main outcome will be postoperative otorrhea as indicated by the Merchant grading scale.

ELIGIBILITY:
Inclusion Criteria:

* Old canal wall down cavity
* Operated between 2011 and 2022

Exclusion Criteria:

* Middle ear cholesteatoma
* Previous obliteration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients operated in our hospital between 2011 and 2022 for troublesome radical cavities that received secondary obliteration
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Number or participants with a dry ear pre- and postoperatively | At 1, 3 and 5-year postoperatively.
  Postoperative otorrhea as indicated by the Merchant grading system. Grade 0-1 was defined as control of infection and grade 2-3 was defined as failure.

SECONDARY OUTCOMES:
Pre- and postoperative air conduction | pre-operatively, in the first 6 months following surgery and 6-12 months postoperatively
  Audiological outcomes pre-operatively, compared to early postoperatively (<6months) and late postoperatively (>6months). Evaluated in the audiometry is the air conduction in decibel.
Pre- and postoperative air-bone gap | pre-operatively, in the first 6 months following surgery and 6-12 months postoperatively
  Audiological outcomes pre-operatively, compared to early postoperatively (<6months) and late postoperatively (>6months). Evaluated in the audiometry is the air-bone gap in decibel.
The number of patients with postoperative surgical complications | First year following surgery
  Complications that occured within the first year following surgery

CONTACTS AND LOCATIONS:
Overall Officials: J.J. Quak, MD, PhD, Principal Investigator — Diakonessenhuis, Utrecht
Locations (1):
- Diakonessenhuis, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided